CLINICAL TRIAL: NCT02957045
Title: Alternative Measurements of Cough Pressure and Effects of Epidural Anaesthesia on Cough Pressure
Acronym: ESPIRATOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Lluís Gallart, Principal Investigator_anesthesiologist, Parc de Salut Mar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ESPIRATOS
Record Dates: First submitted 2016-10-17; First posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Respiratory Physiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cough (Experimental)
  Interventions: Procedure: Cough pressure measurement; Device: Pcough

INTERVENTIONS:
Procedure: Cough pressure measurement
Device: Pcough

SUMMARY:
Pressure generated by cough is an expression of expiratory muscle strength. Cough pressure (Pcough) is usually measured with gastric and/or esophageal catheters, but these are often either inconvenient or uncomfortable for the patient. The aim of this study was to evaluate whether central venous, vesical or rectal catheters could be useful to measure cough pressures as alternative sites to standard esophageal and gastric balloons.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75 years and scheduled for colon cancer surgery were recruited.
* Informed consent signed.

Exclusion Criteria:

Rectal surgery, advanced cancer, abdominal wall disorders, respiratory or neuromuscular illness, body mass index > 30, chronic pain, pregnancy and inability to cough adequately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-08; Primary Completion 2008-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Cough pressure | From baseline until 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Aguilera LG, Gallart L, Alvarez JC, Valles J, Gea J. Rectal, central venous, gastric and bladder pressures versus esophageal pressure for the measurement of cough strength: a prospective clinical comparison. Respir Res. 2018 Oct 1;19(1):191. doi: 10.1186/s12931-018-0897-6. PMID 30285741